CLINICAL TRIAL: NCT05941156
Title: Single-center, Open, One-arm Clinical Study of the Safety and Efficacy of Anti-CD56-CAR T Therapy in Relapsed Refractory NK/T Cell Lymphoma /NK Cell Leukemia
Brief Title: Clinical Study of Anti-CD56-CAR-T in the Treatment of Relapsed/Refractory NK/T Cell Lymphoma /NK Cell Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2023-KL123-01
Record Dates: First submitted 2023-05-17; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Extranodal NK T Cell Lymphoma; NK-Cell Leukemia
Keywords: Anti-CD56 CAR-T
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Leukemia, Large Granular Lymphocytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T Cell Infusion (Experimental): Pretreatment was initiated at -5 days prior to CAR T cell reinfusion, and CAR T cell therapy was performed 2 days after completion of chemotherapy. All patients were pretreated with FC regimen, fludarabine: 30mg/m2×3 days, cyclophosphamide: 750mg/m2×1 day. Anti CD56-CAR T cells were transfused back 2 days after chemotherapy. The freeze-thawed cell product solution is injected back into the body as soon as the patient can accept it. The patient's vital signs should be closely monitored throughout the infusion, and oxygen saturation should be measured at 15-minute intervals before, at the end of, and after infusion, and continue until the patient is stable. 30 to 60 minutes before CAR T cell infusion, patients were given 325 to 650 mg of acetaminophen orally to prevent infusion-related reactions; If fever occurred on the day of CAR T cell infusion, lasted less than 24 hours, and had no other toxicity, it was attributed to the infusion T cell response.
  Interventions: Biological: Anti-CD56 CAR T

INTERVENTIONS:
Biological: Anti-CD56 CAR T — CAR T cells were pretreated at -5 days before retransfusion (FC regimen: fludarabine: 30mg/m2×3 days, cyclophosphamide: 750mg/m2×1 day). Anti CD56-CAR T cells were transfused back to the patient 2 days after the end of chemotherapy. 30 to 60 minutes before CAR T cell infusion, patients were given 325 to 650 mg of acetaminophen orally to prevent infusion-related reactions; If fever occurred on the day of CAR T cell infusion, lasted less than 24 hours, and had no other toxicity, it was attributed to the infusion T cell response.

SUMMARY:
To evaluate the safety and efficacy of anti-CD56-CAR T in the treatment of relapsed refractory NK/T cell lymphoma /NK cell leukemia

DETAILED DESCRIPTION:
Extranodal NK/TCL is an aggressive disease with a poor prognosis and a 5-year survival rate of less than 50%. In the absence of effective treatment, median survival for advanced disease is only 6-12 months. A retrospective review of the International Peripheral T-Cell Lymphoma Project recently reported that the median overall survival of NK/TCL was 7.8 months, corresponding to the worst survival of all T-cell lymphoma entities. Therefore, despite good results in the combination of chemoracal-chemotherapy strategies, autologous bone marrow transplantation, and L-asparagase in the treatment of recurrent cases, NK/TCL remains difficult to cure, and the need for alternative therapeutic strategies has prompted researchers to explore new molecular targets.

Nerve cell adhesion molecule 1 (NCAM-1) -CD56 is a member of the immunoglobulin superfamily and is a biomarker of nerve cell adhesion molecule and NK cell. CD56 is highly expressed in NK/T cell lymphomas, skeletal muscle tumors, and malignancies with neurological or neuroendocrine differentiation. CD56-CAR T cells can kill CD56+ neuroblastoma, glioma, and SCLC tumor cells in vitro coculture, and CD56R-CAR+T cells can inhibit tumor growth in vivo when tested against CD56+ human neuroblastoma xenogeneic and SCLC models. CD56-CAR T cells have also been reported as a safe and effective treatment for refractory/relapsing rhabdomyosarcoma. This indicates that CD56 CAR has a wide clinical application prospect and strong potential therapeutic value as a new CAR T target.

CD56 CAR T cells constructed by our laboratory can produce more precise killing effect on tumor cells by converting the immune checkpoint PD-1 signal. The results showed that CD56 CAR T cells could be prepared effectively and kill NK/ T-cell lymphoma cell line SNK-6 in vitro. Compared with traditional second-generation CAR T cells, CD56-CAR T cells prepared in our laboratory showed better killing effect on SNK-6 cells in vitro. At present, no clinical studies on CD56 CAR T therapy for NK/T cell lymphoma have been reported. Therefore, in this study, CD56 CAR T was used to treat relapsed and refractory NK/T cell lymphoma /NK cell leukemia to observe its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardians voluntarily participate and sign the informed consent;
2. Male or female patients aged 18-70 years (including 18 and 70 years);
3. The patient was diagnosed as NK/T cell lymphoma /NK cell leukemia by pathology or flow cytometry, and currently has no effective treatment options, such as relapse after chemotherapy or hematopoietic stem cell transplantation; Alternatively, patients voluntarily choose to administer anti-CD56-CAR T cells as salvage therapy.
4. The following two categories are included:(1)NK/T cell lymphoma;(2) NK cell leukemia.
5. Subject:

(1)There was no remission or residual lesions after treatment, and HSCT (auto/allo-HSCT) was not suitable; (2)Relapse occurred after CR, and HSCT (auto/allo-HSCT) was not suitable; (3)Patients with high risk factors; (4)Relapse or no remission after hematopoietic stem cell transplantation or cellular immunotherapy.

6. Measurable or evaluable lesions;

7. The patient's main tissues and organs function well:

1. Liver function: ALT/AST < 3 times the upper limit of normal (ULN) and total bilirubin ≤34.2μmol/L;
2. Renal function: creatinine < 220 μmol/L;
3. Lung function: indoor oxygen saturation ≥95%;
4. Cardiac function: left ventricular ejection fraction (LVEF) ≥40%.

8. The patients had not received any anti-cancer treatment such as chemotherapy, radiotherapy, immunotherapy (such as immunosuppressive drugs) within the first 4 weeks of enrollment, and their previous treatment-related toxic reactions had recovered to ≤ grade 1 at the time of enrollment (except low toxicity such as hair loss);

9. The patient's peripheral shallow venous blood flow is smooth, which can meet the needs of intravenous infusion;

10. Patients with ECOG score ≤2 and expected survival time ≥3 months.

Exclusion Criteria:

1. Women who are pregnant (urine/blood pregnancy test positive) or breastfeeding;
2. Men or women who have planned to become pregnant within the last 1 year;
3. The patients were not guaranteed to take effective contraceptive measures (condoms or contraceptives, etc.) within 1 year after enrollment;
4. Patients had uncontrollable infectious diseases within 4 weeks prior to enrollment;
5. Active hepatitis B/C virus;
6. HIV-infected patients;
7. Suffering from a serious autoimmune disease or immunodeficiency disease;
8. The patient is allergic to antibodies, cytokines and other macromolecular biological drugs;
9. The patient had participated in other clinical trials within 6 weeks prior to enrollment;
10. Systemic use of hormones within 4 weeks prior to enrollment (except for inhaled hormones);
11. Suffers from mental illness;
12. The patient has substance abuse/addiction;
13. According to the researchers' judgment, the patient had other conditions that were not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From 1 month to 1 year.
  CR+PR.1.Leukemia:Complete Response (CR):Bone marrow blast cells <5%; primitive cells without Auer bodies; without extramedullary leukemia;Absolute blood neutrophil count was> 1.0*10^9 / L (1000 / μ L);Platelet count> 100*10^9 / L (100 000 / μ L);Not dependent on RBC infusion.Partial Response (PR):Only for Phase I and II clinical trials;Bone marrow cells were reduced to 5 - 25% and at least 50% compared with before treatment;Hematological parameters met the same criteria for CR. 2.Lymphoma:CR:All the evidence of the lesions disappeared.PR:The lymph nodes shrank with no new lesions.
progression-free survival (PFS) | From 1 month to 1 year.
  The time between treatment and observation of disease progression or death from any cause.
overall survival (OS) | From 1 month to 1 year.
  The time from the start of treatment to death from any cause.
event-free survival (EFS) | From 1 month to 1 year.
  The time between the start of treatment and the occurrence of any event, including disease recurrence, death, and so on.
Safety evaluation index | From 1 month to 1 year.
  1. Detection of CRS-related factors: such as IFN, IL-6, TNF, IL-10, IL-4, CRP, etc;2. Testing of various laboratory items: blood routine, coagulation function, blood film observation, liver function, renal work, electrolytes, blood glucose, cardiac enzymes, blood cells, T cell subsets, immunoglobulins, etc;3.Adverse events and serious adverse events were observed.

SECONDARY OUTCOMES:
CAR T cell index of correlation | From 1 month to 1 year.
  The presence of peripheral blood and bone marrow CAR-T cells were measured regularly by using flow cytometry, quantitative PCR techniques.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No